## An eHealth intervention to increase depression treatment initiation and adherence among veterans referred for mental health services (CDA 18-189)

NCT05990075

November 30, 2022

## Analysis plan:

Data processing. Data will be checked for out of range values and missing data where appropriate through plotting and descriptive analyses. Finally, data will be transformed as needed to create the variables of interest (e.g. age of depression onset as age of first episode visible in the EHR). Missing Data Strategies. We will minimize the level of missing data (due to loss to follow-up, withdrawal, or missing assessments) to the extent possible. If missing data occur, I will assess the missing data mechanism for data missing due to loss to follow-up or withdrawal. I will compare baseline measures (e.g., demographics, clinical history, etc.) between subjects that have complete outcome data and those that do not using logistic regression. Multiple imputation will be used for missing data in conjunction with a pattern of missingness. Missing data will be evaluated on an ongoing basis and recruitment may be continued beyond the original sample to achieve the desired power for the proposed analyses. Data Analysis. First, descriptive analyses will be performed on all baseline patient characteristics extracted for all patients approached for study enrollment, including those who agreed and did not agree to participate. To compare these two groups, we will use student t-tests (for continuous variables) and chi-square analysis (for categorical variables). This information will be used to derive acceptability of the proposed intervention. Next, descriptive analyses will be performed on the baseline questionnaires collected from the group of participants enrolled. This will give us additional data about patient characteristics that may further refine our phenotypes or improve study feasibility in the future. Feasibility will be derived from percentage of prompts completed per days of participation in the intervention. Finally, we will calculate rates of treatment initiation (and corresponding 95% confidence interval) and compare to the initiation rate identified in the literature. To compare study treatment initiation to rates we will calculate the 95% confidence interval (CI) for the difference score between proportions (see Franklin, 2007). A significant difference will be denoted if the 95% CI does not include zero (Cumming & Finch, 2005).